CLINICAL TRIAL: NCT05987436
Title: Effects of Supervised Versus Unsupervised Aerobic Exercise Training on Weight Loss, Functional Capacity, Quality of Life and Depression Level in Patients With Essential Hypertension
Brief Title: Effect of Aerobic Exercise in Patients With Essential Hypertension
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Hasan Kara, Medical Doctor, TC Erciyes University
Other Study IDs: HKara2
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Aerobic Exercise; Essential Hypertension
Keywords: supervised aerobic exercise; functional capacity; quality of life; depression level; essential hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group 1 exercised for six weeks, involving once per day, five sessions per week under the supervision of a medical doctor, and a nurse in the aerobic exercise laboratory. The aerobic exercise training program lasted six weeks, and patients lived in the hospital for the whole period. Aerobic exercise training was performed on cycle ergometers (Ergoline, ergoselect II 100/200/Reha, Germany) equipped with a computed ergometer and developed to monitor electrocardiography (ECG), heart rhythm, and BP. Each session consisted of a 5-minute warm-up, followed by 50 minutes of aerobic exercise with an intensity of 50% to 70% of heart rate reserve, calculated by Karvonen formula, and ended with a 5-min cool-down period.
  Interventions: Other: Supervised Aerobic Exercise
- Group 2: The subjects assigned to the control group (Group 2) were advised to maintain dietary habits and physical activity levels and the aerobic exercise program was provided to them after completing the study.

INTERVENTIONS:
Other: Supervised Aerobic Exercise — Group 1 exercised for six weeks, five sessions per week under the supervision of a medical doctor in the aerobic exercise laboratory.
  Groups: Group 1

SUMMARY:
The goal of this observational study is to evaluate the effects of a supervised aerobic exercise training program on weight loss, functional capacity, quality of life (QoL), and depression levels in patients with essential hypertension.

DETAILED DESCRIPTION:
Patients who chose the treatment type according to personal preferences were divided into two groups: Group 1(n:91) exercised for six weeks, five sessions per week under the supervision of a medical doctor in the aerobic exercise laboratory, and group 2(n:47) was advised to maintain dietary habits and physical activity levels. Body weight, serum lipid levels, functional capacity, QoL, and depression level of all the participants were evaluated at baseline and 6 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Absence of concomitant other metabolic and cardiovascular diseases.

Exclusion Criteria:

* Having suffered an event of ischaemic heart disease (<6 months),
* Secondary hypertension,
* Hypertrophic obstructive cardiomyopathy,
* Congestive heart failure,
* Uncontrolled cardiac arrhythmia,
* Thyroid dysfunction,
* Diabetes mellitus,
* Symptomatic peripheral arterial occlusive disease,
* Aortic insufficiency or stenosis,
* Pulmonary or heart disease with dyspnoea at small or moderate effort,
* An outbreak of orthopedic problems on hip, knee or ankles, such as arthroplasty, contracture or severe osteoarthritis,
* Using of antidepressant or anxiolytic drugs,
* Pregnancy,
* Cognitive disfunction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Essential Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Body weight | was measured at the pre-treatment period and the post-treatment 6th week for all the participants by the same physician.
  kilograms
Blood samples | Twelve-hour fasting blood samples were collected between 6.00 am, and 10.00 am at baseline and week 6.
  Serum total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, very-low-density lipoprotein (VLDL) cholesterol, and triglycerides
The functional capacity | 6MWT was assessed in face-to-face interviews before and immediately after the treatment was completed.
  The 6MWT test and the estimated metabolic equivalents or METs were used performed to evaluate functional capacity.
Quality of Life | SF36 was assessed in face-to-face interviews before and immediately after the treatment was completed.
  Quality of life was assessed with Short Form-36 (SF-36).
Depression level | BDI was assessed in face-to-face interviews before and immediately after the treatment was completed.
  Depression level was assessed Beck Depression Inventory (BDI).

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Faculty of Medicine, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No